CLINICAL TRIAL: NCT06964958
Title: LASER - a Phase 2 Trial of 177Lu-PSMA-617 as Systemic Therapy for Renal Cell Carcinoma
Acronym: LASER
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Praful Ravi, MB BCHir, MRCP, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-216
Record Dates: First submitted 2025-05-07; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Renal Cell Carcinoma; Advanced Clear Cell Renal Cell Carcinoma; Kidney Cancer
Keywords: Renal Cell Carcinoma; Advanced Clear Cell Renal Cell Carcinoma; Kidney Cancer; ccRCC; Prostate-specific membrane antigen; PSMA
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Pluvicto

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental: 177Lu-PSMA-617 (Experimental): Enrolled participants will complete:
  * Baseline visit
    --Imaging every 12 weeks, or 2 cycles
  * Cycles 1 through 2:
    * Day 1: Predetermined dose of 177Lu-PSMA-617 1x daily
    * PSMA PET scan before Cycle 3 Day 1
  * Cycles 3 through 6:
    --Day 1: Predetermined dose of 177Lu-PSMA-617 1x daily
  * End of treatment visit with assessments
  * Follow Up: every 6 months for up to 5 years
  * If no radiographic responses of Complete or Partial Response are seen in the first 9 participants enrolled, the trial will terminate. If 1 or more responses are seen in the first 9 participants, the study will enroll an additional 15 participants.
  Interventions: Drug: 177Lu-PSMA-617

INTERVENTIONS:
Drug: 177Lu-PSMA-617 — A radioligand therapy, single-dose vial, via intravenous (into the vein) infusion per protocol.
  Other Names: Pluvicto; Lutetium Lu 177 vipivotide tetraxetan

SUMMARY:
This study aims to evaluate the efficacy and safety of 177Lu-PSMA-617 as a systemic therapy in patients with PSMA-positive advanced clear cell renal cell carcinoma (ccRCC).

The name of the study drug involved in this research study is:

-177Lu-PSMA-617 (a type of radioligand therapy)

DETAILED DESCRIPTION:
The goal of this single-center, phase 2 research study is to evaluate the efficacy and safety of 177Lu-PSMA-617 as a systemic therapy in participants with PSMA-positive advanced clear cell renal cell carcinoma (ccRCC). 177Lu-PSMA-617 aims to deliver targeted radiation to cancer cells, leading to cell death.

The U.S. Food and Drug Administration (FDA) has not approved 177Lu-PSMA-617 as a treatment option for advanced ccRCC, but the study drug is approved for advanced prostate cancer.

The research study procedures include screening for eligibility, in-clinic visits, blood tests, Computerized Tomography (CT) scans, Magnetic Resonance Imaging (MRI) scans, and Prostate-Specific Membrane Antigen Positron Emission Tomography (PSMA PET) scans.

Participants will receive study treatment for up to 6 cycles, or approximately 252 days, and will be followed every 6 months for up to 5 years after discontinuing treatment.

It is expected that about 24 people will take part in this research study.

Novartis Pharmaceuticals Corporation is supporting this research study by supplying the study drug (177Lu-PSMA-617) and providing funding for the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced or metastatic renal cell carcinoma with a clear cell component. Patients with sarcomatoid histology are eligible.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm (≥2 cm) by chest x-ray or as ≥10 mm (≥1 cm) with CT scan, MRI, or calipers by clinical exam. See Section 12 (Measurement of Effect) for the evaluation of measurable disease.
* Age ≥18 years.
* Prior receipt of at least one immune checkpoint inhibitor and at least one tyrosine kinase inhibitor in the neoadjuvant, adjuvant or metastatic settings. Prior treatment with Ra-223 is permitted providing that the last dose was ≥90 days prior to study entry.
* Presence of ≥1 PSMA-avid lesion (with uptake > liver) on baseline/screening 68Ga-PSMA-11 PSMA-PET/CT (within 28 days of planned C1D1), and the absence of any measurable PSMA-negative lesions (i.e. nodal, soft tissue or visceral lesions >1cm) on baseline/screening 68Ga-PSMA-11 PSMA-PET. All patients considered for the study should have their PSMA-PET imaging reviewed in a multidisciplinary meeting with Medical Oncology and Nuclear Medicine to confirm eligibility.
* ECOG performance status ≤2.
* Adequate organ and marrow function as per the below table:

  * System Laboratory Value
  * Hematologic

    * ANC ≥ 1.5×109/L
    * Platelets ≥100×109/L
    * Hemoglobin ≥9g/dL (≥90g/L), independent of transfusions
  * Hepatic

    * Total bilirubin ≤1.5 × ULN OR <2 × ULN if known or suspected Gilbert's syndrome
    * ALT and AST ≤3 × ULN OR ≤5 × ULN if liver metastases present
  * Renal ---eGFR ≥50 mL/min/1.73 m2 (based on Cockcroft-Gault formula OR 24 hour urine collection
* The effects of 177Lu-PSMA-617 on the developing human fetus are unknown. For this reason and because radiopharmaceutical therapies are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Female partners of child-bearing potential should also use highly effective birth control methods throughout the male participant's study treatment and for at least 14 weeks following the last dose of 177Lu-PSMA-617. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and at least 14 weeks following the last dose of 177Lu-PSMA-617.
* Ability to understand and the willingness to sign a written informed consent document. (Providing consents in as many languages as possible is encouraged)

Exclusion Criteria:

* Prior PSMA-targeted therapy (eg. 177Lu-PSMA-617).
* Participants who have had radiotherapy within 4 weeks prior to planned cycle 1 day 1 of study treatment.
* Participants who have received anti-neoplastic intervention or experimental anti-neoplastic therapy within 14 days of planned cycle 1 day 1 of study therapy.
* Participants who are receiving any other investigational agents.
* Participants with untreated brain metastases. Participants with treated brain metastases are eligible if follow-up brain imaging at least 4 weeks after central nervous system (CNS)-directed therapy shows no evidence of progression and ongoing corticosteroids are not required. Participants with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy.
* Participants who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia. Sensory neuropathy grade ≤2 is acceptable.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 177Lu-PSMA-617.
* Symptomatic cord compression, or clinical or radiologic findings indicative of impending cord compression.
* Concurrent active malignancy whose natural history or treatment has the potential to interfere with safety or efficacy assessment of the investigational regimen. Patients with non-melanomatous skin cancer, superficial bladder cancer, cancer not needing active therapy for at least 2 years, cancer for which the treating investigator deems the subject to be in remission, or any prior malignancy that was treated with curative intent (no evidence of disease for at least 3 years) are permitted to enroll.

NB - participants who are found to have suspected prostate cancer on the basis of PSMA-PET/CT performed for screening (eg. PSMA avid disease in the prostate) are eligible to proceed on study on the basis of clinical judgement by the treating physician. Prostate (or other) biopsy is not required to confirm evidence of prostate cancer, if suspected, prior to proceeding with study therapy as long as the treating physician deems RCC to be a more pressing treatment priority.

* The participant has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
* Females that are pregnant and/or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Tumor assessment will be performed every 12 weeks on treatment. Treatment duration is 36 weeks.
  ORR is defined as the proportion of participants who experienced complete response (CR) or partial response (PR) during treatment. Tumors will be assessed for response and progression by RECIST version 1.1 by central radiology review.

SECONDARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | Adverse events are collected every study visit until the discontinuation of treatment plus 30 days. Treatment duration is 36 weeks.
  Adverse events will be graded and analyzed using CTCAE v5.
Median Disease-free Survival (DFS) | Tumor assessment will be performed every 12 weeks on treatment. Treatment duration is 36 weeks.
  Disease-free survival (PFS) is defined as the time from the date of treatment initiation to the earlier of progression or death due to any cause. Participants alive without disease are censored at date of last disease evaluation.
Median Overall Survival (OS) | Survival follow-up will be every 6 months until 5 years after discontinuing treatment. The treatment duration is 36 weeks.
  OS is Overall survival based on the Kaplan-Meier method is defined as the time from randomization to death. Participants alive are censored at the last date of contact (including lost-to-follow-up) or at the date of withdrawal of consent, if relevant.

CONTACTS AND LOCATIONS:
Overall Officials: Praful Ravi, MB BCHir, MRCP, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu